CLINICAL TRIAL: NCT06065306
Title: Potential Diagnostic Biomarkers for Aortic Dissection in the Emergency Department: the Aggrecan, Desmosine, D-dimer-Emergency Department (ADD-ED) Study
Brief Title: Potential Diagnostic Biomarkers for Aortic Dissection in the Emergency Department
Acronym: ADD-ED
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: CREC 2022.631
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Aortic Dissection
Keywords: aortic dissection; biomarker; diagnostic; d-dimer; aggrecan; desmosine
MeSH Terms: conditions — Aortic Dissection; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AD: Patient aged greater than 18, presented to the ED with first 24 hours of symptoms suggesting AD, including chest pain, upper back pain, syncope of unknown cause, symptoms of any acute perfusion deficit and confirmed AD.
- Healthy: Patients attending ED who do not have coronary disease, hypertension or aortic disease would be identified as healthy control.

SUMMARY:
The goal of this observational study is to determine the utility of desmosine, D-dimer and aggrecan as early diagnostic biomarkers in aortic dissection. The main questions it aims to answer are:

* To investigate the plasma levels of selected biomarkers in ED patients with confirmed aortic dissection
* To study the diagnostic performance of plasma levels of selected biomarkers for aortic dissection
* To study the association between plasma levels of selected biomarkers and clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presentation to the ED with first 24 hours of symptoms suggesting AD, including chest pain, upper back pain, syncope of unknown cause, symptoms of any acute perfusion deficit
* Confirmed AD

  * the diagnosis of AD adjudicated by an independent expert panel at hospital discharge or death, whichever comes first
  * The expert panel will consist of (1) a specialist in Emergency Medicine and (2) a specialist in Cardiology and (3) a specialist in Cardiothoracic Surgery.

Exclusion Criteria:

* Age <18 years old
* Pregnancy
* Surgery or stenting performed before recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or above, with AD presenting to the ED within the first 24 hours of symptom onset will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum levels of D-Dimer, Aggrecan and Desmosine | Blood samples taken preoperatively
  Biomarkers :Serum levels of D-Dimer, Aggrecan and Desmosine will be compared in patients with confirmed AD versus age and sex matched healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided